CLINICAL TRIAL: NCT02553226
Title: Continued Versus Discontinued Oxytocin Stimulation of Labour in a Double-blind Randomised Controlled Trial
Brief Title: Continued Versus Discontinued Oxytocin Stimulation of Labour
Acronym: CONDISOX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Randers Regional Hospital (Other); Aarhus University Hospital (Other); Kolding Sygehus (Other); Aalborg University Hospital (Other); Herning Hospital (Other); Rigshospitalet, Denmark (Other); University of Amsterdam (Other); Hillerod Hospital, Denmark (Other); Odense University Hospital (Other); Hvidovre University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 01102015
Record Dates: First submitted 2015-06-28; First posted 2015-09-17 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2019-09

CONDITIONS: Adverse Reaction to Oxytocin
Keywords: Active phase of labour; Discontinuation; Caesarean section
MeSH Terms: interventions — Oxytocin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continued group (Active Comparator): Recieve routine treatment with oxytocin according to the danish national guidelines.
  Interventions: Drug: Oxytocin
- discontinued group (placebo) (Placebo Comparator): The routine treatment with oxytocin will be discontinued and replaced with isotonic saline, when the active phase of labour is established.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — Both arms will initially receive routine treatment with oxytocin according to national guidelines. When active phase of labour is established both arms will have their infusion-set changed for a blinded infusion-set.
  Other Names: syntocinon
  Arms: Continued group
Drug: Placebo — Both arms will initially receive routine treatment with oxytocin according to national guidelines. When active phase of labour is established both arms will have their infusion-set changed for a blinded infusion-set.
  Other Names: Isotonic saline
  Arms: discontinued group (placebo)

SUMMARY:
Background:

The proposed study will investigate the effect of Syntocinon® (synthetic oxytocin) to induce labour. The hypothesis to be studied is that once the active phase of labour has commenced, Syntocinon® can be discontinued and the labour process will continue.

Design:

Double-blind randomised controlled multicentre trial

Setting:

Aarhus University Hospital, Denmark and Regional Hospital of Randers, Denmark

Population:

1200 women (600 in each group) stimulated in the latent phase of labour with oxytocin for induction

Methods:

The Syntocinon® infusion will be replaced with either continuous isotonic saline (placebo) or Syntocinon® infusion (control group), when the active phase of labour is reached.

Main outcome measures:

Caesarean section (primary outcome), tachysystole, neonatal asphyxia, birth experience

Perspective:

Syntocinon® is on the list high-alert medications and associated with complications for mother and child during labour. Reducing the duration of stimulation during labour may lower the number of asphyxial sequelae and the number of caesarean sections.

DETAILED DESCRIPTION:
Randomisation:

When the orificium ≥6 cm, regular painful contractions (≥3 per 10 minutes) and rupture of membranes participants will be randomised in a 1:1 ratio to either the control (continued Syntocinon®) or intervention (discontinued Syntocinon®) group using an Internet-based randomisation programme. The randomisation can only be performed when the woman consents to participation. Written consent can be given after the commencement of the Syntocinon® infusion, provided the woman previously has received sufficient information for her to give properly informed consent. Random block-sizes of 8 are used, and the participants will be stratified by site (Aarhus University Hospital, Randers Regional Hospital, Aalborg University hospital, or Sygehus Lillebælt Kolding), parity (nulliparous or parous) and indication for Syntocinon® infusion (induction or induction due to premature rupture of membranes).

The randomisation number corresponds to number of the project medicine (ampoule). The personnel of the delivery ward will administer the ampoules according to existing guidelines concerning medicine administration

Oxytocin stimulation protocol:

Existing national procedures prior to stimulation will be followed, including use of the existing checklists. No further examination will be done prior to inclusion and stimulation, no blood samples nor ECG to identify e.g. unknown QT-syndrome will be performed as this is never performed as a standard procedure prior to induction.

Latent phase: Stimulation will be given according to national DSOG guidelines7. Initially 20 ml/hour of 10 IE Syntocinon® diluted in 1000 ml 0,9% NaCl. The dose rate will be increased every 20 minutes by 20 ml/hour until appropriate uterine activity of 3-5 contractions per 10 minutes is achieved. The maximum allowed dose rate 180 ml/hour for induction of labour.

Active phase: The woman will be included in the study, when the active phase of labour is established (cervical dilatation ≥ 6 cm, ≥3 contractions per 10 minutes, and rupture of membranes). Randomisation is performed, and the infusion will be replaced by the trial solution, which will be either Syntocinon® at the same concentration, or a placebo infusion which will not contain Syntocinon®:

1. Control group; 10 IE Syntocinon® diluted in 1000 ml 0,9% NaCl infusion
2. Intervention group; 1ml 0,9% NaCl diluted in 1000ml 0,9% NaCl infusion. The infusion will be continued to achieve uterine activity of 3-5 contractions per 10 minutes. Maximum allowed dose is 180 ml/hour for induction. The procedure for administration of the trial solution is identical with the existing procedure.

Complications:

The infusion will be reduced or discontinued at any point of labour, if the following occur:

* Hyperstimulation (>5 contractions per 10 minutes and non-reassuring CTG13). A management algorithm for this situation is made.
* Uterine contractions lasting 2 minutes or more
* Non-reassuring CTG (recurrent variable decelerations, fetal tachycardia or bradycardia, minimal to absent baseline variability, late decelerations)
* Suspicion of uterine rupture These conditions will be managed according to the guidelines of the local delivery wards.

Dystocia:

If there is failure to progress, defined as less than two cm dilation over 4 hours despite apparently adequate contractions and/or maximal infusion rates (Syntocinon® or placebo), the project medicine will be replaced with open-labelled Syntocinon® infusion. Stimulation will be given according to national DSOG guidelines7. Initially 20 ml/hour of 10 IE Syntocinon® diluted in 1000 ml 0,9% NaCl. The dose rate will be increased every 20 minutes by 20 ml/hour until appropriate uterine activity of 3-5 contractions per 10 minutes is achieved. The maximum allowed dose rate is180 ml/hour for induction.

Woman receiving open-labelled Syntocinon® infusion for 4 hours and continuous failure to progress: Consider caesarean section.

Unconcealment The primary investigator or a nominated deputy will at all time be able to break the randomisation code and reveal the allocation group, if needed. The Internet Based Randomisation Programme will provide the primary investigator or a nominated deputy with this possibility. (A 24/7 availability of the allocation group is thereby provided).

Side effects and risks:

Persistent failure to progress can be expected in 8-46% of the participants in the placebo group versus 3-17% in the control group. 3 4 5 6 Based on data from the pilot study, the risk of caesarean section is expected to be 15% in the placebo group versus 22% in the control group. According to the pilot study and previous studies 3 4 5 6, the maternal and neonatal complications in the placebo group are expected to be lower than in the control group.

All participants are monitored with continuous electronic fetal heart rate monitoring during labour to detect complications such as uterine tachysystole and non-reassuring/pathological fetal heart rate, in accordance with national guidelines.

The personnel of the delivery ward are responsible for registering of adverse reactions and adverse events.

Following adverse reactions and event will be registered immediately in the electronic medical journal of the patient:

* Cesarean delivery
* Postpartum hemorrhage >500 ml
* Manual placenta removal
* Rupture of the anale sphincter
* Urine retention
* Neonatal: pH <7,10 and/or Apgar score ≤ 6 at 5 minutes

Following serious adverse reactions and adverse events will be also registered immediately in the electronic medical journal of the patient:

* Intrauterine dead during labour
* Maternal amniotic fluid emboli or thromboembolic event
* Maternal cardiac arrest
* Maternal Pulmonary edema
* Uterine rupture The women will be followed for at least 3-6 hours postpartum (termination of project medicine) according current practice on the delivery ward.

The product resume of Syntocinon® will be used as reference to determine whether a Serious Adverse Reaction is expected or unexpected. Primary investigator or a nominated deputy will go through the participants medical file 7-30 days postpartum during data management and Primary investigator will ensure that all relevant information about suspected serious unexpected adverse reactions that are fatal or life-threatening is recorded and reported as soon as possible to the competent authorities concerned, and to the Ethics Committee, and in any case no later than seven days after the knowledge such a case, and that relevant follow-up information is subsequently communicated within an additional eight days.

Primary investigator will report to the competent authorities concerned and to the Ethics Committee concerned all other suspected unexpected serious adverse reactions as soon as possible but within a maximum of 15 days of first knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Women stimulated with Syntocinon® infusion for induction of labour (with or without cervical priming by prostaglandin)

Exclusion Criteria:

* Unable to read and understand the Danish language or to give informed consent
* Cervical dilatation > 4 cm
* Non-cephalic presentation
* Multiple gestation
* Pathological fetal heart rate pattern (cardiotocogram, CTG) before Syntocinon® initiation
* Fetal weight estimation > 4500 g (clinical or ultrasonic)
* Subject declines participation
* Gestational age less than 37 completed weeks

Definition: Stimulation with Syntocinon® following Premature Rupture of membranes (PROM) is induction of labour if there is no cervical change prior to starting the infusion, whereas stimulation with Syntocinon after PROM but following the establishment of significant cervical change is augmentation.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2016-04; Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Caesarean section | labour
  Frequency of acute performed caesarean sections

SECONDARY OUTCOMES:
Instrumental delivery | 0-48 hours
  use of vacuum extraction or forceps for delivery
Birth experience | 4 weeks postpartum
  Childbirth Experience Questionaire (CEQ)
Breastfeeding | 0-6months
  Time to established feeding and duration of exclusive breastfeeding.
Duration of the active phase of labour | 0-48 hours
  Maternal outcome
Total duration of labour | 0-48 hours
  (from initiation time of stimulation with Syntocinon until delivery)
Uterine tachysystoli | 0-48 hours
  Parturition will be monitored with continous CTG
Uterine hyperstimulation | 0-48 hours
  Parturition will be monitored with continous CTG
Use of epidural analgesia | 0-48 hours
Dose and duration of oxytocin infusion | 0-48 hours
Use of episiotomy | 0-48 hours
Rupture of the anal sphincter | 0-48 hours
Uterine rupture | 0-48 hours
Volume of blood loss at delivery and postpartum | 0-48 hours
Need for evacuation of retained products of conception | 0-48 hours
Maternal use of antibiotics during labour | 0-48 hours
Maternal readmission | 0-168 hours
Retention of urine | 0-48 hours
  requiring catheterisation
Vaginal explorations | 0-48 hours
  number
Cardiotocogram (CTG) classification | 0-48 hours
  Parturition will be monitored with continous CTG. Suspicious, pathologic or terminal CTG will be registered.
Fetal scalp pH values or Fetal scalp lactate | 0-48 hours
Apgar score at 1 and 5 minutes | 0-48 hours
Umbilical cord arterial pH | 0-48 hours
Neonatal use of antibiotics - postpartum | 0-48 hours
Neonatal hyperbilirubinaemia | 0-48 hours
  High values of bilirubinaemi, which leads to treatment, will be registered
Neonatal admission | 0-48 hours
  Admission in Neonatal Intensive Care Unit (NICU)
Need for resuscitation/ventilation of the newborn | 0-48 hours
  (bag, mask, CPAP, and/or intubation, time to onset of spontaneous ventilation)
Neonatal death | 0-7 days
Time of birth of placenta | 0-2 hours
Cause of maternal readmission | 0-7 days
  Suspected infection, Endometritis proven with culture, Urinary tract infection treated with antibiotics, Wound infection treated with abtibiotics, Bowel obstruction, Pneumonia, Trombo-embolic complications, Eclampsia, HELLP, Admission due to child, no maternal reason

CONTACTS AND LOCATIONS:
Overall Officials: Niels Uldbjerg, DMSc, Principal Investigator — Aarhus University Hospital; Pinar Bor, PhD, Principal Investigator — Regionalhospital Randers; Julie Glavind, PhD, Principal Investigator — Regionalhospital Randers; Philip Steer, BSc, Principal Investigator — Imperial College, London, England
Locations (10):
- Denmark (9):
  - Aarhus University Hospital, Aarhus, Aarhus N
  - Aalborg University Hospital, Aalborg
  - Rigshospitalet, Copenhagen
  - Regionshospitalet Herning, Herning
  - Nordsjællandshospital, Hillerød
  - Hvidovre Hospital, Hvidovre
  - Sygehus LIllebælt, Kolding
  - Odense University Hospital, Odense
  - Department of Gynecology and Obstetrics, Randers
- Academic Medical Center, Amsterdam, Amsterdam-Zuidoost, Netherlands

IPD SHARING:
Plan to Share IPD: No
The trial is GCP monitored by the GCP unit of Aarhus University Hospital, Odense University Hospital, Copenhagen University and The GCP unit at the AMC
  Members of the Data Monitoring Committee:
  Chair: Lone Krebs (Obstetrician) Member: Gorm Greisen (Pediatrician) Member: Martin Johansen (Statistician)
  Members of the Trial Steering Committee:
  Chair: Jim Thornton Member: Thomas bergholt Member: Jens Fuglsang Member: Wessel Ganzevoort

REFERENCES:
- [Derived] Boie S, Glavind J, Uldbjerg N, Steer PJ, Bor P; CONDISOX trial group. Continued versus discontinued oxytocin stimulation in the active phase of labour (CONDISOX): double blind randomised controlled trial. BMJ. 2021 Apr 14;373:n716. doi: 10.1136/bmj.n716. PMID 33853878
- [Derived] Boie S, Glavind J, Uldbjerg N, Bakker JJH, van der Post JAM, Steer PJ, Bor P. CONDISOX- continued versus discontinued oxytocin stimulation of induced labour in a double-blind randomised controlled trial. BMC Pregnancy Childbirth. 2019 Sep 2;19(1):320. doi: 10.1186/s12884-019-2461-x. PMID 31477047